CLINICAL TRIAL: NCT04122508
Title: Are Dental Neglect and the Presence of Siblings Risk Factors for Oral Health in Children
Brief Title: Are Dental Neglect and the Siblings Risk Factors in Children
Status: Completed | Type: Observational
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Sema Aydınoglu, assistant professor, Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: 62
Record Dates: First submitted 2019-10-05; First posted 2019-10-10 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Behavior, Child; Caries,Dental; Neglect, Child; Anxiety
Keywords: anxiety; siblings; dental caries; oral health; child abuse
MeSH Terms: conditions — Child Behavior; Dental Caries; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Neglect insidiously affects a child's overall health in all aspects. The aim of this study was to determine whether the presence of siblings caused dental neglect, and whether there was a relationship between dental neglect and anxiety.

DETAILED DESCRIPTION:
Dental neglect is an intentional failure of parents or caregivers to take precautions and fulfil necessary dental treatment, and has a close relationship with dental caries and anxiety. Oral health status of the children was evaluated using the DMFT/dmft, PUFA/pufa, and OHI-S indices. In addition, the parents completed the Dental Neglect Scale (DNS) and a questionnaire, and the Modified Child Dental Anxiety Scale (MCDASf) was administered to the children to assess their dental anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 6 and 12 years old
* Being healthy
* Being volunteer for the study

Exclusion Criteria:

* Systemic and mental disorders
* Syndromes or other major health diseases
* Cooperation problems

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: children who presented for the first time to the Faculty of Dentistry in Rize
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
the effects of presence of siblings on dental neglect | for eight months from the beginning of the study
  The effects of presence of siblings on oral health and dental neglect was assessed using dental neglect scale. The dental neglect scale for children was originally composed of seven statements, using a Likert scale ranging from one to five . The total score of DNS can range from 7 to 35, with higher scores representing greater dental neglect.
the effects of presence of siblings on oral health | for eight months from the beginning of the study
  the effects of presence of siblings on oral health and dental neglect was assessed using oral hygiene index . The OHI-S has two elements, the Debris Index and the Calculus Index. The Debris Index and the Calculus Index can range from 0 to 3, the oral hygiene index values from 0 to 6.
the effects of presence of siblings on dental caries | for eight months from the beginning of the study
  the effects of presence of siblings on oral health and dental neglect was assessed using, DMFT/dmft index. caries (D/d), missing due to caries (M/m), filling (F/f) teeth were recorded using DMF-T indices for permanent teeth and dmf-t indices for primary teeth.
the effects of presence of siblings on untreated caries | for eight months from the beginning of the study
  the effects of presence of siblings on oral health and dental neglect was assessed using pufa index. The index recorded the presence of visible pulp involvement (P/p), mucosal ulceration due to root fragments (U/u), fistulae (F/f) and/or abscessess (A/a). Higher scores represents worse oral health.

SECONDARY OUTCOMES:
to evaluate whether there was a correlation between dental neglect and anxiety in children | for eight months from the beginning of the study
  the relationship between dental neglect and anxiety was evaluated using Modified Child Dental Anxiety Scale (MCDASf). MCDASf, which is a validated and reliable indicator for the measurement of dental anxiety in children was used. Children in this study were asked to complete the MCDASf, which covers eight multiple choice statements with five faces ranging from 1 (not anxious), to 5 (extremely anxious). The total score on the MCDASf was calculated for each subject (ranging from 5: little or no dental anxiety, to 40: severe dental anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Sema Aydınoglu, Dr, Principal Investigator — Recep Tayyip Erdogan University Training and Research Hospital
Locations (1):
- Recep Tayyip Erdogan University Training and Research Hospital, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available 5 years after publication
Access Criteria: Data access requests will be reviewed by authors.